CLINICAL TRIAL: NCT00343460
Title: A Pivotal Phase 3 Observer-Blind, Randomized Clinical Trial of the Efficacy and Safety of APF530 Compared to Aloxi For The Prevention of Acute-Onset and Delayed-Onset Chemotherapy-Induced Nausea and Vomiting Following The Administration of Either Moderately or Highly Emetogenic Chemotherapy Regimens
Brief Title: APF530 or Aloxi (Palonosetron Hydrochloride) Combined With Dexamethasone in Preventing Nausea and Vomiting in Patients Receiving Chemotherapy for Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Heron Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: C2006-01; APPA-C2006-01
Record Dates: First submitted 2006-06-22; First posted 2006-06-23 (Estimated); Results first posted 2016-12-28 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Nausea and Vomiting; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: nausea and vomiting; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Nausea; Vomiting | interventions — Granisetron; Dexamethasone; Palonosetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm I (Active Comparator): Patients receive palonosetron hydrochloride IV, placebo subcutaneously (SC), and dexamethasone IV on day 1 of chemotherapy course 1. Patients in the high-risk (level 5) stratum also receive oral dexamethasone on days 2-4 of all treatment courses.
  Interventions: Drug: dexamethasone; Drug: Palonosetron Hydrochloride; Other: placebo
- Arm II (Experimental): Patients receive APF530 SC, placebo IV, and dexamethasone IV on day 1 of chemotherapy course 1. Patients then receive APF530 SC and dexamethasone IV on day 1 of chemotherapy courses 2-4. Patients in the high-risk (level 5) stratum also receive oral dexamethasone as in arm I.
  Interventions: Drug: APF530; Drug: dexamethasone; Other: placebo
- Arm III (Experimental): Patients receive APF530 SC at a higher dose, placebo IV, and dexamethasone IV on day 1 of chemotherapy course 1. Patients then receive APF530 SC (at the same higher dose) and dexamethasone IV on day 1 of chemotherapy courses 2-4. Patients in the high-risk (level 5) stratum also receive oral dexamethasone as in arm I.
  Interventions: Drug: APF530; Drug: dexamethasone; Other: placebo

INTERVENTIONS:
Drug: APF530 — Given subcutanously
  Arms: Arm II; Arm III
Drug: dexamethasone — Given IV and orally
Drug: Palonosetron Hydrochloride — Given IV
  Arms: Arm I
Other: placebo — Given subcutanously or IV

SUMMARY:
This randomized phase III trial is studying APF530 and dexamethasone to see how well they work compared with palonosetron and dexamethasone in preventing nausea and vomiting in patients receiving chemotherapy for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the overall activity and effects of APF530 versus palonosetron hydrochloride in combination with dexamethasone for prophylaxis of acute- or delayed-onset, chemotherapy-induced nausea and vomiting in patients undergoing moderately or highly emetogenic chemotherapy for cancer.

Secondary

* Evaluate the safety, tolerability, and efficacy of APF530, in terms of prevention of acute- and delayed-onset nausea and vomiting, in these patients.
* Gather the pharmacokinetics of APF530 in a subset of patients during chemotherapy course 1.
* Gather ECG data (using 24-hour Holter monitoring) in a subset of patients during chemotherapy course 1.

OUTLINE: This is a randomized, placebo-controlled, double-blind, parallel-group, multicenter study. Patients are stratified according to emetogenicity of scheduled chemotherapy (moderate-risk [level 3 or 4] vs high-risk [level 5]). Patients are randomized to 1 of 3 treatment arms (I, II, and III). Patients who are randomized to receive palonosetron hydrochloride during chemotherapy course 1 (arm I) are then re-randomized to 1 of 2 treatment arms (II and III) after chemotherapy course 1 to receive treatment during chemotherapy courses 2-4.

Patients receive palonosetron hydrochloride or APF530 and/or placebo 30-60 minutes before the start of chemotherapy. Patients receive dexamethasone 30-90 minutes before the start of chemotherapy.

* Arm I: Patients receive palonosetron hydrochloride IV, placebo subcutaneously (SC), and dexamethasone IV on day 1 of chemotherapy course 1. Patients in the high-risk (level 5) stratum also receive oral dexamethasone on days 2-4 of all treatment courses.
* Arm II: Patients receive APF530 SC, placebo IV, and dexamethasone IV on day 1 of chemotherapy course 1. Patients then receive APF530 SC and dexamethasone IV on day 1 of chemotherapy courses 2-4. Patients in the high-risk (level 5) stratum also receive oral dexamethasone as in arm I.
* Arm III: Patients receive APF530 SC at a higher dose, placebo IV, and dexamethasone IV on day 1 of chemotherapy course 1. Patients then receive APF530 SC (at the same higher dose) and dexamethasone IV on day 1 of chemotherapy courses 2-4. Patients in the high-risk (level 5) stratum also receive oral dexamethasone as in arm I.

A subset of patients undergo blood collection periodically during study for analysis of plasma APF530 concentration.

Quality of life is assessed on day 5 after completion of chemotherapy course 1.

After completion of study treatment, patients are followed at approximately 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed malignant disease

  * No head and neck cancer or upper gastrointestinal cancer
* Scheduled to receive a single day of moderately or highly emetogenic chemotherapy regimen (for ≤ 4 courses)

  * Chemotherapy administration ≤ 4 hours
  * Duration of each course ≤ 28 days
  * Causing nausea and vomiting in 30-100% of patients if untreated according to Hesketh algorithm
* Must be able to receive standardized doses of dexamethasone for the prevention of emesis during study treatment
* No greater than mild nausea or any vomiting within 24 hours before beginning study treatment

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known allergy or hypersensitivity to other selective 5-HT3 receptor antagonists or local anesthetics
* QTc interval ≤ 500 ms
* No cardiac abnormality predisposing the patient to arrhythmia
* No psychological problem that, in the opinion of the investigator, is severe enough to preclude study participation
* No recent history (i.e., ≤ 1 year) of alcohol or drug abuse
* No concurrent condition that, in the opinion of the investigator, could affect assessment of study medication or interfere with the nausea/vomiting response (e.g., severe renal or hepatic impairment)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No radiotherapy 7 days prior to, during, and 5 days after completion of study treatment
* More than 7 days since prior chemotherapy
* More than 7 days since prior and no concurrent prohibited medications (e.g., CYP3A4 inhibitors or other antiemetic medications)
* More than 7 days since prior antinausea medications
* More than 30 days since prior treatment on an investigational trial
* No other concurrent corticosteroids or dexamethasone at a different dose than study treatment
* No concurrent use of APF530, palonosetron hydrochloride, or aprepitant as rescue medications

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1428 (Actual)
Dates: Start 2006-06; Primary Completion 2008-09 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Barr, PhD, Study Chair — Heron Therapeutics
Locations (52):
- United States (52):
  - Anniston Oncology, PC, Anniston, Alabama
  - Palo Verde Hematology Oncology - Glendale, Glendale, Arizona
  - Arizona Clinical Research Center, Incorporated, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Pacific Cancer Medical Center, Incorporated, Anaheim, California
  - Southbay Oncology / Hematology Medical Group, Campbell, California
  - Compassionate Cancer Care Medical Group Incorporated - Corona, Corona, California
  - Compassionate Cancer Care Medical Group Incorporated - Fountain Valley, Fountain Valley, California
  - Advanced Research Management Services, Incorporated, Los Angeles, California
  - Kenmar Research Institute, Los Angeles, California
  - Medical Oncology Care Associates - Orange, Orange, California
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Providence Hospital, Washington D.C., District of Columbia
  - Pasco Pinellas Cancer Center - New Port Richey, New Port Richey, Florida
  - Innovative Medical Research of South Florida, Incorporated, North Miami Beach, Florida
  - Columbus Clinic, PC, Columbus, Georgia
  - Clintell, Incorporated, Skokie, Illinois
  - Investigative Clinical Research, LLC, Indianapolis, Indiana
  - Cancer Center of Indiana, New Albany, Indiana
  - Family Medicine of Vincennes Clinical Trial Center, Vincennes, Indiana
  - Medical Center Vincennes, Vincennes, Indiana
  - Kentucky Cancer Clinic - Hazard, Hazard, Kentucky
  - Kentuckiana Cancer Institute, PLLC, Louisville, Kentucky
  - Hematology-Medical Oncology Associates at Central Maine Comprehensive Cancer Center, Lewiston, Maine
  - Mercy Medical Center, Baltimore, Maryland
  - Center for Cancer and Blood Disorders at Suburban Hospital, Bethesda, Maryland
  - Center for Clinical Research at Washington County Hospital, Hagerstown, Maryland
  - Northern Michigan Hospital, Petoskey, Michigan
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Kansas City Cancer Centers - South, Kansas City, Missouri
  - Star Hematology & Oncology, Phillipsburg, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Falck Cancer Center at Arnot Ogden Medical Center, Elmira, New York
  - Hudson Valley Hematology-Oncology Associates - Poughkeepsie, Poughkeepsie, New York
  - Comprehensive Cancer Center at Pardee Hospital, Hendersonville, North Carolina
  - Boice Willis Clinic, PA, Rocky Mount, North Carolina
  - Eastern North Carolina Medical Group, PLLC, Rocky Mount, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Gabrail Cancer Center - Canton Office, Canton, Ohio
  - Gabrail Cancer Center - Dover Office, Dover, Ohio
  - MedCentral - Mansfield Hospital, Mansfield, Ohio
  - Signal Point Hematology Oncology Incorporated, Middletown, Ohio
  - Cancer Treatment Centers of America at Southwestern Regional Medical Center, Tulsa, Oklahoma
  - Pottsville Cancer Clinic, Pottsville, Pennsylvania
  - Charleston Hematology Oncology Associates, PA, Charleston, South Carolina
  - Julie and Ben Rogers Cancer Institute at Memorial Hermann Baptist Beaumont Hospital, Beaumont, Texas
  - Texas Cancer Clinic, San Antonio, Texas
  - Cancer Outreach Associates - Abingdon, Abingdon, Virginia
  - Virginia Oncology Care, PC, Richlands, Virginia
  - Western Washington Oncology, Incorporated, PS at Western Washington Cancer Center, Lacey, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boccia R, O'Boyle E, Cooper W. Randomized phase III trial of APF530 versus palonosetron in the prevention of chemotherapy-induced nausea and vomiting in a subset of patients with breast cancer receiving moderately or highly emetogenic chemotherapy. BMC Cancer. 2016 Feb 26;16:166. doi: 10.1186/s12885-016-2186-4. PMID 26921245
- [Derived] Raftopoulos H, Boccia R, Cooper W, O'Boyle E, Gralla RJ. Slow-release granisetron (APF530) versus palonosetron for chemotherapy-induced nausea/vomiting: analysis by American Society of Clinical Oncology emetogenicity criteria. Future Oncol. 2015 Sep;11(18):2541-51. doi: 10.2217/fon.15.185. Epub 2015 Aug 20. PMID 26289588

RESULTS

PARTICIPANT FLOW:
Groups:
- APF530 5 mg: APF530 5 mg - Safety Population
- APF530 10 mg: APF530 10 mg - Safety Population
- Aloxi 0.25 mg: Aloxi 0.25 mg - Safety Population
Period: Cycle 1
Arm/Group | APF530 5 mg | APF530 10 mg | Aloxi 0.25 mg
Started | 475 | 481 | 472
Completed | 453 | 459 | 454
Not Completed | 22 | 22 | 18
Period: Cycle 2 - 4
Arm/Group | APF530 5 mg | APF530 10 mg | Aloxi 0.25 mg
Started | 584 | 565 | 0
Completed | 528 | 515 | 0
Not Completed | 56 | 50 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat Population
Groups:
- Cycle 1 APF530 5 mg - Moderately; Cycle 1 APF530 10 mg - Moderately; Cycle 1 Aloxi 0.25 mg - Moderately: Cycle 1 - Modified Intent-to-Treat Population
  Emetogenic Status: Moderately
- Cycle 1 APF530 5 mg - Highly; Cycle 1 APF530 10 mg - Highly; Cycle 1 Aloxi 0.25 Highly: Cycle 1 - Modified Intent-to-Treat Population
  Emetogenic Status: Highly
- Total: Total of all reporting groups
Arm/Group | Cycle 1 APF530 5 mg - Moderately | Cycle 1 APF530 10 mg - Moderately | Cycle 1 Aloxi 0.25 mg - Moderately | Cycle 1 APF530 5 mg - Highly | Cycle 1 APF530 10 mg - Highly | Cycle 1 Aloxi 0.25 Highly | Total
Number analyzed (Participants) | 214 | 212 | 208 | 229 | 240 | 238 | 1341
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (12.80) | 55.1 (12.79) | 57.3 (12.36) | 57.6 (13.35) | 56.8 (13.20) | 58.1 (13.74) | 56.62 (13.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189 | 177 | 177 | 153 | 152 | 158 | 1006
  Male | 25 | 35 | 31 | 76 | 88 | 80 | 335

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Complete Response (CR) During Acute Phase (0-24 Hours) After Administration of Chemotherapy Course 1
Description: Complete Response is defined as no emetic episodes and no use of rescue medications
Time Frame: 0-24 Hours
Population: Cycle 1 - Modified Intent-to-Treat Population
Measure: Number; unit: participants
Arm/Group | Cycle 1 APF530 5 mg - Moderately | Cycle 1 APF530 10 mg - Moderately | Cycle 1 Aloxi 0.25 mg - Moderately | Cycle 1 APF530 5 mg - Highly | Cycle 1 APF530 10 mg - Highly | Cycle 1 Aloxi 0.25 Highly
Number analyzed (Participants) | 214 | 212 | 208 | 229 | 240 | 238
participants | 160 | 163 | 156 | 178 | 195 | 192

2. Primary Outcome: Proportion of Patients With CR During Delayed-onset Phase (24-120 Hours) After Administration of Chemotherapy Course 1
Description: Complete Response is defined as no emetic episodes and no use of rescue medications
Time Frame: 24-120 Hours
Population: Cycle 1 - Modified Intent-to-Treat Population
Measure: Number; unit: participants
Arm/Group | Cycle 1 APF530 5 mg - Moderately | Cycle 1 APF530 10 mg - Moderately | Cycle 1 Aloxi 0.25 mg - Moderately | Cycle 1 APF530 5 mg - Highly | Cycle 1 APF530 10 mg - Highly | Cycle 1 Aloxi 0.25 Highly
Number analyzed (Participants) | 214 | 212 | 208 | 229 | 240 | 238
participants | 110 | 125 | 120 | 148 | 164 | 158

3. Secondary Outcome: Proportion of Patients With Complete Control During the Acute Phase (0-24 Hours), Delayed-onset Phase (24-120 Hours), and During Chemotherapy Course 1
Description: Complete control is defined as complete response with no more than mild nausea.
Time Frame: 0-120 Hours
Population: Cycle 1 - Modified Intent-to-Treat Population
Measure: Number; unit: participants
Arm/Group | Cycle 1 APF530 5 mg - Moderately | Cycle 1 APF530 10 mg - Moderately | Cycle 1 Aloxi 0.25 mg - Moderately | Cycle 1 APF530 5 mg - Highly | Cycle 1 APF530 10 mg - Highly | Cycle 1 Aloxi 0.25 Highly
Number analyzed (Participants) | 214 | 212 | 208 | 229 | 240 | 238
participants
  CC during acute Phase | 154 | 152 | 147 | 170 | 183 | 184
  CC during the delayed-onset phase | 100 | 115 | 107 | 138 | 150 | 147
  CC during the overall risk period | 93 | 107 | 99 | 127 | 138 | 136

4. Secondary Outcome: Proportion of Patients With Total Response During the Acute Phase, Delayed-onset Phase, and During Chemotherapy Course 1
Description: TR during acute phase is defined as Complete Response with no nausea during 0 to 24 hours following the administration of chemotherapy in Cycle 1.
  TR during delayed-onset phase is defined as Complete Response with no nausea during >24 to 120 hours following the administration of chemotherapy in Cycle 1. TR during overall risk period is defined as Complete Response with no nausea during 0 to 120 hours following the administration of chemotherapy in Cycle 1.
Time Frame: 0-120 Hours
Population: Cycle 1 - Modified Intent-to-Treat Population
Measure: Number; unit: participants
Arm/Group | Cycle 1 APF530 5 mg - Moderately | Cycle 1 APF530 10 mg - Moderately | Cycle 1 Aloxi 0.25 mg - Moderately | Cycle 1 APF530 5 mg - Highly | Cycle 1 APF530 10 mg - Highly | Cycle 1 Aloxi 0.25 Highly
Number analyzed (Participants) | 214 | 212 | 208 | 229 | 240 | 238
participants
  TR during acute phase | 135 | 121 | 113 | 141 | 146 | 158
  TR during the delayed-onset phase | 76 | 89 | 73 | 115 | 113 | 122
  TR during the overall risk period | 68 | 79 | 65 | 103 | 101 | 117

5. Secondary Outcome: Number of Emetic Episodes
Description: Number of Emetic Episodes - days 1-5
Time Frame: Days 1-5
Population: Cycle 1 - Modified Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: Number of Emetic Episodes
Arm/Group | Cycle 1 APF530 5 mg - Moderately | Cycle 1 APF530 10 mg - Moderately | Cycle 1 Aloxi 0.25 mg - Moderately | Cycle 1 APF530 5 mg - Highly | Cycle 1 APF530 10 mg - Highly | Cycle 1 Aloxi 0.25 Highly
Number analyzed (Participants) | 208 | 208 | 205 | 217 | 236 | 222
Number of Emetic Episodes | 3.4 (8.03) | 3.1 (9.35) | 2.1 (5.12) | 2.3 (6.69) | 2.4 (7.87) | 2.5 (7.15)

6. Secondary Outcome: Time to First Treatment Failure
Description: Proportions of subjects event free at 24, 48, 72, 96, and 120 hours after chemotherapy administration
Time Frame: 0-120 Hours
Population: Proportions of subjects event free in Cycle 1 - Modified Intent-to-Treat Population
Measure: Number; unit: Proportion of subjects event free
Groups:
- Cycle 1 Aloxi 0.25 - Highly: Cycle 1 - Modified Intent-to-Treat Population
  Emetogenic Status: Highly
Arm/Group | Cycle 1 APF530 5 mg - Moderately | Cycle 1 APF530 10 mg - Moderately | Cycle 1 Aloxi 0.25 mg - Moderately | Cycle 1 APF530 5 mg - Highly | Cycle 1 APF530 10 mg - Highly | Cycle 1 Aloxi 0.25 - Highly
Number analyzed (Participants) | 214 | 211 | 208 | 228 | 238 | 238
Proportion of subjects event free
  24 Hours | 0.738 | 0.763 | 0.755 | 0.781 | 0.811 | 0.803
  48 Hours | 0.636 | 0.659 | 0.635 | 0.706 | 0.723 | 0.714
  72 Hours | 0.533 | 0.564 | 0.567 | 0.649 | 0.685 | 0.672
  96 Hours | 0.485 | 0.550 | 0.534 | 0.618 | 0.668 | 0.634
  120 Hours | 0.485 | 0.540 | 0.529 | 0.600 | 0.647 | 0.620

7. Secondary Outcome: First and Overall Use of Rescue Medication
Time Frame: 0-120 Hours
Population: Cycle 1 - Modified Intent-to-Treat Population
Measure: Number; unit: participants
Arm/Group | Cycle 1 APF530 5 mg - Moderately | Cycle 1 APF530 10 mg - Moderately | Cycle 1 Aloxi 0.25 mg - Moderately | Cycle 1 APF530 5 mg - Highly | Cycle 1 APF530 10 mg - Highly | Cycle 1 Aloxi 0.25 - Highly
Number analyzed (Participants) | 214 | 212 | 208 | 229 | 240 | 238
participants
  Used Rescue Medication, 0-24 hours | 42 | 37 | 41 | 35 | 23 | 25
  Used Rescue Medication, 24-120 hours | 83 | 69 | 63 | 60 | 42 | 42
  Used Rescue Medication, 0-120 hours | 89 | 76 | 72 | 71 | 45 | 49

8. Secondary Outcome: Severity of Nausea Daily and During Chemotherapy Course 1 (0-120 Hours)
Description: Maximum severity of nausea, days 1-5
Time Frame: 0-120 Hours
Population: Severity of Nausea - Cycle 1 - Modified Intent-to-Treat Population
Measure: Number; unit: participants
Arm/Group | Cycle 1 APF530 5 mg - Moderately | Cycle 1 APF530 10 mg - Moderately | Cycle 1 Aloxi 0.25 mg - Moderately | Cycle 1 APF530 5 mg - Highly | Cycle 1 APF530 10 mg - Highly | Cycle 1 Aloxi 0.25 - Highly
Number analyzed (Participants) | 212 | 210 | 204 | 219 | 235 | 232
participants
  None | 78 | 85 | 66 | 105 | 102 | 121
  Mild | 45 | 53 | 68 | 53 | 68 | 53
  Moderate | 59 | 40 | 46 | 48 | 37 | 39
  Severe | 30 | 32 | 24 | 13 | 28 | 19

9. Secondary Outcome: Sustainability of Antiemetic Effect of APF530 Over Multiple Chemotherapy Courses
Description: Sustainability of Overall Complete Response (CR 0-120 hrs) Over Two, Three, and Four Cycles
  Complete Response is defined as no emetic episodes and no use of rescue medications
Time Frame: 0-120 Hours
Population: Number of subjects in the Modified Intent-to-Treat Population with overall CR (0-120 hrs) in all cycles
Measure: Number; unit: participants with overall CR
Groups:
- Cycles 1, 2, 3 and 4 - Moderately; Cycles 1, 2, 3 and 4 - Highly: APF530 5 mg
- Cycles 1, 2, 3, and 4 - Moderately; Cycles 1, 2, 3, and 4 - Highly: APF530 10 mg
Arm/Group | Cycles 1, 2, 3 and 4 - Moderately | Cycles 1, 2, 3, and 4 - Moderately | Cycles 1, 2, 3 and 4 - Highly | Cycles 1, 2, 3, and 4 - Highly
Number analyzed (Participants) | 91 | 92 | 106 | 95
participants with overall CR | 34 | 35 | 56 | 52

10. Secondary Outcome: Quality of Life and the Impact of Nausea and Vomiting on Day 5
Description: Functional Living Index
Time Frame: 5 days
Population: Cycle 1 - Modified Intent-to-Treat Population (All Languages Except Punjabi)
Measure: Number; unit: participants
Arm/Group | Cycle 1 APF530 5 mg - Moderately | Cycle 1 APF530 10 mg - Moderately | Cycle 1 Aloxi 0.25 mg - Moderately | Cycle 1 APF530 5 mg - Highly | Cycle 1 APF530 10 mg - Highly | Cycle 1 Aloxi 0.25 - Highly
Number analyzed (Participants) | 208 | 210 | 204 | 223 | 228 | 231
participants
  No nausea impact on daily life | 112 | 127 | 120 | 142 | 142 | 159
  No vomiting impact on daily life | 157 | 162 | 160 | 173 | 182 | 191

11. Secondary Outcome: Patient's Global Satisfaction With Antiemetic Therapy During Acute Phase and Chemotherapy Course 1
Description: Subject who were very satisfied on Day 1
Time Frame: 0- 24 Hours
Population: Cycle 1 - Modified Intent-to-Treat Population
Measure: Number; unit: participants
Arm/Group | Cycle 1 APF530 5 mg - Moderately | Cycle 1 APF530 10 mg - Moderately | Cycle 1 Aloxi 0.25 mg - Moderately | Cycle 1 APF530 5 mg - Highly | Cycle 1 APF530 10 mg - Highly | Cycle 1 Aloxi 0.25 - Highly
Number analyzed (Participants) | 211 | 212 | 208 | 229 | 240 | 238
participants | 101 | 113 | 98 | 128 | 128 | 135

ADVERSE EVENTS:
Groups:
- Cycle 1 APF530 5 mg; Cycle 1 APF530 10 mg; Cycle 1 Aloxi 0.25 mg: Serious Treatment-Emergent Adverse Events - Cycle 1 - Safety Population
- Cycles 2-4 APF530 5 mg; Cycle 2-4 APF530 10 mg: Serious Treatment-Emergent Adverse Events - Cycles 2-4 - Safety Population
Arm/Group | Cycle 1 APF530 5 mg | Cycle 1 APF530 10 mg | Cycle 1 Aloxi 0.25 mg | Cycles 2-4 APF530 5 mg | Cycle 2-4 APF530 10 mg
Serious Adverse Events (participants affected / at risk) | 42/464 | 36/468 | 27/472 | 61/528 | 73/515
Other Adverse Events (participants affected / at risk) | 335/464 | 349/468 | 313/472 | 422/528 | 413/515
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cycle 1 APF530 5 mg (N=464) | Cycle 1 APF530 10 mg (N=468) | Cycle 1 Aloxi 0.25 mg (N=472) | Cycles 2-4 APF530 5 mg (N=528) | Cycle 2-4 APF530 10 mg (N=515)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 6 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 7 | 3 | 5 | 8
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 2 | 2 | 6
Pancytopenia (Blood and lymphatic system disorders) | 2 | 2 | 1 | 2 | 2
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1 | 0 | 1 | 3
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Sudden Death (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Diabetes mellitus (Endocrine disorders) | 1 | 0 | 1 | 1 | 0
Hyperglycaemia (Endocrine disorders) | 0 | 1 | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 2
Diverticulitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 3 | 2 | 3 | 1
Oesophageal carcinoma recurrent (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 4 | 1 | 1 | 3
Asthenia (General disorders) | 0 | 1 | 0 | 1 | 1
Chest pain (General disorders) | 1 | 1 | 1 | 1 | 2
Death (General disorders) | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (General disorders) | 1 | 0 | 0 | 1 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 3 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bronchitis chronic (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Catheter related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 7 | 4
Respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 2 | 4 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 2 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Prothrombin level abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 2 | 4 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Bladder cancer (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 2 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 4 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 6
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 4 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Appendicectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Mastectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 1
Tumour excision (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Vascular disorders) | 0 | 0 | 1 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 1 | 0 | 4 | 3
Epistaxis (Vascular disorders) | 1 | 0 | 0 | 1 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 3 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Septic phlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cycle 1 APF530 5 mg (N=464) | Cycle 1 APF530 10 mg (N=468) | Cycle 1 Aloxi 0.25 mg (N=472) | Cycles 2-4 APF530 5 mg (N=528) | Cycle 2-4 APF530 10 mg (N=515)
Anaemia (Blood and lymphatic system disorders) | 46 | 42 | 34 | 86 | 87
Neutropenia (Blood and lymphatic system disorders) | 39 | 48 | 38 | 46 | 42
Thrombocytopenia (Blood and lymphatic system disorders) | 18 | 16 | 13 | 32 | 36
Abdominal pain (Gastrointestinal disorders) | 21 | 13 | 28 | 15 | 24
Constipation (Gastrointestinal disorders) | 61 | 72 | 62 | 78 | 79
Diarrhoea (Gastrointestinal disorders) | 47 | 44 | 39 | 51 | 69
Dyspepsia (Gastrointestinal disorders) | 16 | 16 | 16 | 32 | 30
Nausea (Gastrointestinal disorders) | 55 | 58 | 41 | 66 | 73
Vomiting (Gastrointestinal disorders) | 24 | 18 | 13 | 28 | 25
Asthenia (General disorders) | 23 | 21 | 30 | 60 | 39
Fatigue (General disorders) | 62 | 62 | 52 | 80 | 94
Injection site bruising (General disorders) | 78 | 93 | 41 | 124 | 153
Injection site erythema (General disorders) | 33 | 51 | 14 | 58 | 61
Injection site haemorrhage (General disorders) | 20 | 18 | 10 | 35 | 31
Injection site nodule (General disorders) | 22 | 50 | 3 | 57 | 90
Injection site pain (General disorders) | 16 | 33 | 5 | 34 | 37
Oedema peripheral (General disorders) | 13 | 7 | 8 | 28 | 31
Pyrexia (General disorders) | 15 | 15 | 19 | 32 | 24
Upper respiratory tract infection (Infections and infestations) | 4 | 4 | 9 | 29 | 21
Decreased appetite (Metabolism and nutrition disorders) | 13 | 17 | 17 | 24 | 32
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 11 | 10 | 35 | 29
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 10 | 10 | 29 | 21
Dizziness (Nervous system disorders) | 14 | 17 | 8 | 21 | 29
Headache (Nervous system disorders) | 31 | 47 | 44 | 38 | 44
Insomnia (Nervous system disorders) | 20 | 25 | 11 | 27 | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 11 | 14 | 31 | 34
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 12 | 9 | 35 | 19
Alopecia (Skin and subcutaneous tissue disorders) | 19 | 31 | 25 | 82 | 69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A period of 60 working days for presentational material and abstracts and 90 days for manuscripts is permitted for the sponsor's review. The sponsor can request modifications of any manuscript or other materials to be published or presented. The sponsor can also request additional time to obtain additional patent protection or take such other measures to establish and preserve its intellectual property and proprietary rights before publishing information from this trial.